CLINICAL TRIAL: NCT02502357
Title: The Power of Healing Statements on Post Operative Pain Control: A Randomized Controlled Trial
Brief Title: Healing Statements and Their Effect on Post Operative Pain
Acronym: PHSPOPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-043
Record Dates: First submitted 2015-06-16; First posted 2015-07-20 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: pain control; healing statements; pelvic prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: simple randomization
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healing Statements (Experimental): Patients in the healing statements group will be read healing statements during anesthesia induction, prior to undergoing surgery.
  Interventions: Other: Healing Statements
- No Healing Statements (No Intervention): Patients in the no healing statements group will not be read healing statements during anesthesia induction prior to undergoing surgery. They will receive standard of care.

INTERVENTIONS:
Other: Healing Statements — Before the patient in the experimental group is placed under general anesthesia, the study staff member will repeat 5 times:
  "Following this operation, [the participant] will feel very comfortable and [the participant] will heal very well."
  Toward the end of the surgery, the study staff member will say 5 times:
  "The operation has gone very well." "Following the operation, [the participant] will be hungry. [The participant] will be thirsty and urinate easily."
  Arms: Healing Statements

SUMMARY:
This is a randomized clinical trial comparing the severity of post-operative pain and use of pain medication in women who are and are not exposed to healing statements before undergoing vaginal hysterectomy with minimally invasive sacrocolpopexy. The investigators' hypothesis is that those who are read healing statements before surgery will require less post-operative pain medications and experience less severe pain than those who do not hear the statements.

DETAILED DESCRIPTION:
This is a randomized controlled trial of women undergoing vaginal hysterectomy with minimally invasive sacrocolpopexy. Eligible patients will be approached for study participation after they have decided to proceed with the vaginal hysterectomy with minimally invasive sacrocolpopexy. After enrollment, demographics including age, race, prolapse stage, and medical history will be collected. Before vaginal hysterectomy with minimally invasive sacrocolpopexy in the OR, they will be randomized to the group that will be read healing statements or to the group without healing statements. Women randomized to the healing statement group will have the following statements read to them by a trained research staff member, using Peggy Huddleston's technique. Before the patient is placed under general anesthesia, the study staff member will repeat 5 times:

"Following this operation, [the participant] will feel very comfortable and [the participant] will heal very well"

Toward the end of the surgery, the study staff member will say 5 times:

"The operation has gone very well." "Following the operation, [the participant] will be hungry. [The participant] will be thirsty and urinate easily."

Prior to reading these statements to the patient, the research staff member will listen to a previously recorded audio sample of how the statements should be read with regard to tone of voice and attitude.

Patients will then fill out the VAS pain scale 6 and 24 hours after surgery. Pain medication use, dosage, type of medication will be assessed by examining electronic medical records. Time to pass void trial and time to first bowel movement will be recorded on paper and brought to the patient's 2-week follow up visit. Nausea will be assessed 6 and 24 hours after surgery using the Postoperative Nausea and Vomiting (PONV) Intensity Scale. Patients will be given standard post-operative instructions for a vaginal hysterectomy with minimally invasive sacrocolpopexy, and be told to come to the clinic in 2 weeks for a follow up visit. During this time, the will be told to keep a daily diary of pain medication use including name, dosage, and amount taken. At the 2-week visit, the patient will fill out another VAS pain scale and PFDI-20 and their pain medication diaries will be collected. The patient's overall sense of recovery will be assessed using the PGI. Once the data is collected, statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo vaginal hysterectomy with minimally invasive sacrocolpopexy
* Age ≥18 years
* English speaking
* Available for 2 week follow up
* Able to complete study questionnaires

Exclusion Criteria:

* History of chronic pain prior to surgery
* Pain during intercourse or in lower abdomen or genital region at baseline prior to index surgery (identified if patient answers yes to question 20 on the Pelvic Floor Distress Inventory-20)
* Hearing impairment
* Pregnancy by self-report or positive pregnancy test
* Active pelvic infection, herpes, candidiasis
* Indication for surgery is due to neoplasm
* History of pain syndromes including fibromyalgia, interstitial cystitis, dysmenorrhea, and depression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
Baseline Pain (analyzed by VAS Numeric Pain Distress Scale) | baseline
  Pain
Post Operative Pain (analyzed by VAS Numeric Pain Distress Scale) | 6 hours after surgery
  Pain
Post Operative Pain (analyzed by VAS Numeric Pain Distress Scale) | 24 hours after surgery
  Pain
Post Operative Pain (analyzed by VAS Numeric Pain Distress Scale) | 2 weeks after surgery
  Pain

SECONDARY OUTCOMES:
Post operative Nausea and Vomiting (analyzed by Post-Operative Nausea and Vomiting Intensity Scale) | 6 hours after surgery and 24 hours after surgery
  Nausea and Vomiting
Time to First Bowel Movement | Followed for 2 weeks after surgery
  Bowel Movement
Time to Pass Void Trial (Urination) | Followed for 2 weeks after surgery
  Urination
Patient Perception of Improvement | 2 weeks after surgery
  Patient Perception of Improvement measured by Patient Global Perception of Improvement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Iglesia, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Evans C, Richardson PH. Improved recovery and reduced postoperative stay after therapeutic suggestions during general anaesthesia. Lancet. 1988 Aug 27;2(8609):491-3. doi: 10.1016/s0140-6736(88)90131-6. PMID 2900410
- [Result] Block RI, Ghoneim MM, Sum Ping ST, Ali MA. Efficacy of therapeutic suggestions for improved postoperative recovery presented during general anesthesia. Anesthesiology. 1991 Nov;75(5):746-55. doi: 10.1097/00000542-199111000-00005. PMID 1952199
- [Result] Liu WH, Standen PJ, Aitkenhead AR. Therapeutic suggestions during general anaesthesia in patients undergoing hysterectomy. Br J Anaesth. 1992 Mar;68(3):277-81. doi: 10.1093/bja/68.3.277. PMID 1547052
- [Result] McLintock TT, Aitken H, Downie CF, Kenny GN. Postoperative analgesic requirements in patients exposed to positive intraoperative suggestions. BMJ. 1990 Oct 6;301(6755):788-90. doi: 10.1136/bmj.301.6755.788. PMID 2224266
- [Result] Huddleston P. Prepare for Surgery, Heal Faster: A Guide of Mindy-Body Techniques. Angel River Press, 2012.
- [Result] Watters M, Feldman J, Schoetz D, Abrams M, Goy C, Catman M, Huddleston P. The Power of Relaxation: A Holistic Approach to Preoperative Patient Education.
- [Result] Huddleston M, Bierbaum B. Cost-effectiveness of Using Mind-Body Techniques for Total Knee-Joint Replacement.
- [Result] Hutchings DD. The value of suggestion given under anesthesia: A report and evaluation of 200 cases. American Journal of Clinical Hypnosis 1961; 26-29.
- [Result] Furlong M. Positive suggestions presented during anaesthesia. Memory and Awareness in Anaesthesia (Amsterdam: Swets & Zeitlinger, 1990).
- [Result] Lebovits AH, Twersky R, McEwan B. Intraoperative therapeutic suggestions in day-case surgery: are there benefits for postoperative outcome? Br J Anaesth. 1999 Jun;82(6):861-6. doi: 10.1093/bja/82.6.861. PMID 10562780
- [Result] Wolfe LS, Millet JB. Control of postoperative pain by suggestion under general anesthesia. American Journal of Clinical Hypnosis 1960; 3:109-112.
- [Result] Steinberg ME, Hord AH, Reed B, Sebels PS. Study of the effect of intraoperative analgesia and well-being. Memory and Awareness in Anesthesia (Englewood Cliffs, NJ: Prenctice Hall, 1993).
- [Derived] Shah NM, Andriani LA, Mofidi JL, Ingraham CF, Tefera EA, Iglesia CB. Therapeutic Suggestion in Postoperative Pain Control: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 Jul 1;27(7):409-414. doi: 10.1097/SPV.0000000000000906. PMID 32541300